CLINICAL TRIAL: NCT02100423
Title: A Phase II Study of Curcumin and Vitamin D in Previously Untreated Patients With Early Stage Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Curcumin and Cholecalciferol in Treating Patients With Previously Untreated Stage 0-II Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Paolo Caimi, MD (Other)
Responsible Party: Sponsor-Investigator, Paolo Caimi, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE5913
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Contiguous Stage II Small Lymphocytic Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage I Small Lymphocytic Lymphoma; Stage II Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Curcumin; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (curcumin, cholecalciferol) (Experimental): Patients receive curcumin PO daily on days 1-28 and cholecalciferol PO daily on days 8-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving partial response or better may receive treatment for a total of 2 years.
  Interventions: Drug: curcumin; Dietary Supplement: cholecalciferol; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: curcumin — Given PO
  Other Names: C.I. 75300; C.I. Natural Yellow 3; CU; Diferuloylmethane
Dietary Supplement: cholecalciferol — Given PO
  Other Names: Calciol; Vitamin D3
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies the efficacy (activity), and tolerability of curcumin and cholecalciferol combination in treating patients with previously untreated stage 0-II chronic lymphocytic leukemia or small lymphocytic lymphoma. Curcumin and cholecalciferol may prevent or slow the growth of cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) based on National Cancer Institute-Working Group (NCI-WG) criteria in chronic lymphocytic leukemia (CLL) or the Cheson criteria in small lymphocytic lymphoma (SLL).

SECONDARY OBJECTIVES:

I. To determine the time to first cytotoxic treatment (TFCT), progression free survival (PFS), and overall survival (OS) using this regimen.

OUTLINE:

Patients receive curcumin orally (PO) daily on days 1-28 and cholecalciferol PO daily on days 8-28 of course 1 and days 1-28 of subsequent courses. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving partial response or better may receive treatment for a total of 2 years.

After completion of study treatment, patients are followed up for 30 days and then every 3-6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of CLL based on peripheral blood flow cytometry and/or bone marrow aspiration and biopsy OR diagnosis of SLL based on lymph node or bone marrow biopsy; patients with SLL need to have measurable disease
* Performance status (Eastern Cooperative Oncology Group [ECOG]) 0-2
* Patients must have not received any prior treatment for CLL or SLL
* Patients must be stage 0-II based on Rai staging system; must have no indication for treatment for SLL per NCI-WG criteria
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* Serum creatinine =< 2.0 g/dL or calculated creatinine clearance (CrCl) >= 60mL/min (Cockcroft-Gault method)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal (ULN)
* Bilirubin < 2.0 x ULN, unless subject has Gilbert's disease
* Calcium < 10.1 mg/dL (corrected to serum albumin)
* Females will be either postmenopausal for at least 1 year or surgically sterile for at least 3 months OR females of child-bearing potential must have a negative pregnancy test at screening and agree to take appropriate precautions to avoid pregnancy (double barrier method of birth control or abstinence) from screening through 3 months after the last dose of treatment
* Able to comprehend and willing to sign an Informed Consent Form (ICF)
* Subjects must be off any steroids 7 days prior to the initiation of treatment
* Subjects must be off any curcumin, tumeric, or vitamin D supplements for 14 days prior to the initiation of treatment
* Subjects must be able to take oral medications

Exclusion Criteria:

* Presence of malignancy (other than the one treated in this study) which required systemic treatment within the past 3 years
* Any indication to start treatment for CLL based on NCI-WG criteria
* Prior therapy for CLL/SLL
* Subjects who are pregnant or breast-feeding; breastfeeding should be discontinued if the mother is treated with curcumin
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Hypercalcemia of any cause
  * Untreated hyperparathyroidism
  * Paget's disease of bone
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements as judged by treating physician; subjects receiving antibiotics that are under control may be included in the study
* Inability to take oral medications
* Patients receiving other investigational agent
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to curcumin or vitamin D or other agents used in this study
* Patients on therapeutic anticoagulation, with heparin (or low-molecular weight heparin), warfarin, or a direct thrombin inhibitor as the safety of concurrent administration of curcumin has not been established
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-16 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caimi, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Started | 35
Completed | 29
Not Completed | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 35
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 1
  50-59 years | 17
  60-69 years | 12
  70-79 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Based on NCI-WG (for CLL) and Cheson Criteria (for SLL)
Description: The point estimate of the overall response rate (biologic response rate + complete response [CR] + partial response [PR]) with 95% confidence intervals will be calculated using binomial distribution theory.
  The time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented and assessed
Time Frame: Up to 2 years
Population: Participants enrolled in study
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 35
percentage of participants | 0

2. Secondary Outcome: Time to First Cytotoxic Treatment (TFCT)
Description: TFCT defined as the time from entry onto study until initiation of treatment with cytotoxic agents because of disease progression.
  Kaplan-Meier method and Cox proportional hazard model will be used for the data analysis.
Time Frame: Up to 2 years
Population: Evaluable participants who progressed. Two additional participants were recorded to have progressed but data are missing regarding TFCT and all efforts to retrieve information have been exhausted.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 4
Months | 10.5 [6 to 21]

3. Secondary Outcome: Percent of Participants With Progression Free Survival (PFS)
Description: Percent of participants that reached 2-year survival without disease progression.
  PFS is defined as the time from entry onto study until CLL/SLL progression or death from any cause. National Cancer Institute Working Group (NCI-WG) criteria is used for CLL participants and Cheson Criteria is used for SLL participants
Time Frame: Up to 2 years
Population: Participants enrolled in study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 35
percentage of participants | 57.5 [44.9 to 100]

4. Secondary Outcome: Overall Survival (OS)
Description: Number of participants still alive at 2 years after treatment discontinuation.
Time Frame: Up to 2 years
Population: Participants enrolled on study.
Measure: Number; unit: participants
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 35
participants | 35

5. Secondary Outcome: Duration of Response
Description: Time from achievement of partial response, complete response or biologic response to disease progression
Time Frame: Up to 2 years
Population: No participants analyzed because there was no therapeutic response
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 0

6. Post Hoc Outcome: Median Overall Survival (OS)
Description: Number of participants still alive at 2 years after treatment discontinuation.
Time Frame: Up to 2 years post-treatment
Population: Participants who received the Curcumin and Cholecalciferol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Curcumin, Cholecalciferol)
Number analyzed (Participants) | 35
Participants | 35

ADVERSE EVENTS:
Time Frame: Through study completion, which was an average of 4 years.
Arm/Group | Treatment (Curcumin, Cholecalciferol)
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Curcumin, Cholecalciferol) (N=35)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Curcumin, Cholecalciferol) (N=35)
Anemia (Blood and lymphatic system disorders) | 7 (12)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Intermittent night sweats (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (45)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Stomach cramps (Gastrointestinal disorders) | 1 (1)
Stool color change (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 5 (6)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 14 (17)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 3 (5)
Infection under chin (Infections and infestations) | 1 (1)
Lymph gland infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (5)
Alkaline phosphatase increased (Investigations) | 6 (8)
Aspartate aminotransferase increased (Investigations) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (7)
White blood cell count increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (6)
Lymphocyte count increased (Investigations) | 7 (8)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 9 (13)
Weight gain (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (24)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
low vitamin D level (Metabolism and nutrition disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Night sweats (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Flu like symptoms, body aches (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Brittle nails (Skin and subcutaneous tissue disorders) | 1 (1)
Skin integrity (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Night sweats (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT02100423/Prot_SAP_000.pdf